CLINICAL TRIAL: NCT02410343
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Efficacy, Safety and Tolerability Study of TV-1106 in Growth Hormone-Deficient Adults Who Are Not Current Users of rhGH Treatment
Brief Title: Study of TV-1106 in Growth Hormone-Deficient Adults
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV1106-IMM-30021; 2014-003796-32 (EudraCT Number)
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Growth Hormone Deficiency
Keywords: long acting growth hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — albusomatropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo was injected subcutaneously once weekly on the same day and time for 24 weeks. To maintain the blind, placebo could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 to match the effect of dose titration.
  Interventions: Drug: Placebo
- TV-1106 (Experimental): TV-1106 was injected subcutaneously once weekly on the same day and time for 24 weeks. A common starting dose was 5.0 mg. Doses could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 until the participant's insulin-like growth factor 1 (IGF-1) standard deviation score (SDS) was within the range of -0.5 to +1.5.
  Interventions: Drug: TV-1106

INTERVENTIONS:
Drug: TV-1106 — A starting dose of 5.0 mg was expected to be appropriate for most patients because the daily recommended starting dose of recombinant human growth hormone (rhGH) treatments (e.g. somatropin) is 0.2 mg/day, and the conversion factor was 28. Dosage could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 until the participant's insulin-like growth factor 1 (IGF-1) standard deviation score (SDS) was within the range of -0.5 to +1.5.
  Other Names: long-acting growth hormone, albutropin
  Arms: TV-1106
Drug: Placebo — Placebo treatment was administered in a blinded fashion and titrated on weeks 4, 8, 12 and 16 to mimic the active treatment.
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of 6 months of treatment with TV-1106 compared with placebo on body fat composition.

ELIGIBILITY:
Inclusion:

* males and females 18 years of age or over
* diagnosis of adult growth hormone deficiency (GHD) for at least 6 months, or patients who have hypopituitarism from surgical resection
* no history of exposure to any rhGH within the past 12 months prior to screening
* stable, adequate doses of replacement hormones (adrenal, thyroid, estrogen, testosterone, vasopressin) for at least 3 months prior to screening

  * Other criteria apply, please contact the investigator for more information

Exclusion:

* patients with acute or chronic conditions or diseases that could confound results of the study or put the patient at undue risk as determined by the investigator
* Presence of contraindications to rhGH treatment
* patients who have participated in another clinical trial with a new chemical/biological entity within 3 months of screening
* patients with known active malignancy (excluding surgically removed basal cell carcinoma or carcinoma in situ of cervix)
* patients with a previously treated pituitary tumor with evidence of tumor progression in the past year patients with a new diagnosis of pituitary adenoma or other intracranial tumor within 12 months of screening
* presence of Prader-Willi syndrome, Turner's syndrome, untreated adrenal insufficiency, active acromegaly in the past 5 years, or active Cushing's syndrome in the past 1 year
* patients with type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus as indicated by a glycated hemoglobin (HBA1c) of ≥8%
* patients using weight reducing agents or appetite suppressants
* women who are pregnant or nursing, or planning pregnancy during the study period

  * Other criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (33):
- United States (25):
  - Teva Investigational Site 13102, Artesia, California
  - Teva Investigational Site 13127, Fountain Valley, California
  - Teva Investigational Site 13126, Fountain Valley, California
  - Teva Investigational Site 13103, Miami, Florida
  - Teva Investigational Site 13118, Miami, Florida
  - Teva Investigational Site 13123, Miami, Florida
  - Teva Investigational Site 13492, Miami, Florida
  - Teva Investigational Site 13114, Miami Lakes, Florida
  - Teva Investigational Site 13100, Pembroke Pines, Florida
  - Teva Investigational Site 13121, West Palm Beach, Florida
  - Teva Investigational Site 13104, Chicago, Illinois
  - Teva Investigational Site 13124, Evansville, Indiana
  - Teva Investigational Site 13101, Detroit, Michigan
  - Teva Investigational Site 13112, Henderson, Nevada
  - Teva Investigational Site 13113, Las Vegas, Nevada
  - Teva Investigational Site 13109, Brooklyn, New York
  - Teva Investigational Site 13494, New York, New York
  - Teva Investigational Site 13106, New York, New York
  - Teva Investigational Site 13096, Asheville, North Carolina
  - Teva Investigational Site 13108, Pittsburgh, Pennsylvania
  - Teva Investigational Site 13110, Arlington, Texas
  - Teva Investigational Site 13125, Dallas, Texas
  - Teva Investigational Site 13097, Houston, Texas
  - Teva Investigational Site 13107, Houston, Texas
  - Teva Investigational Site 13120, Houston, Texas
- Teva Investigational Site 33030, Linz, Austria
- Teva Investigational Site 54112, Moravskoslezsky, Czechia
- Greece (2):
  - Teva Investigational Site 63054, Athens
  - Teva Investigational Site 63053, Chaïdári
- Hungary (2):
  - Teva Investigational Site 51197, Budapest
  - Teva Investigational Site 51195, Pécs
- Teva Investigational Site 30112, Brescia, Italy
- Teva Investigational Site 50303, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 46 patients screened, 14 patients at 10 centers located in the US and Europe (Austria, Greece, Hungary) met entry criteria and were considered eligible for randomization. Of the 32 patients not randomly assigned to study treatment, 26 were excluded on the basis of inclusion/exclusion criteria and 6 were excluded for "other" reasons.
Pre-assignment Details: Participants were randomly allocated to 1 of 2 treatment groups (TV-1106 or placebo) in a 2:1 allocation to prevent selection bias.
Groups:
- Placebo: Placebo was injected subcutaneously once weekly on the same day and time for 24 weeks during the Core Period. To maintain the blind, placebo could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 to match the effect of dose titration. Participants who completed the Core Period were eligible to enter an open-label extension phase for 12 additional months where all participants received treatment with TV-1106.
- TV-1106: TV-1106 was injected subcutaneously once weekly on the same day and time for 24 weeks during the Core Period. A common starting dose was 5.0 mg. Doses could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 until the participant's insulin-like growth factor 1 (IGF-1) standard deviation score (SDS) was within the range of -0.5 to +1.5. Participants who completed the Core Period were eligible to enter an open-label extension phase for 12 additional months where all participants received treatment with TV-1106.
Period: Core Period (24 Weeks)
Arm/Group | Placebo | TV-1106
Started | 6 | 8
Completed | 1 | 1
Not Completed | 5 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Early termination of study by sponsor | 4 | 7
Period: Extension Period (12 Months)
Arm/Group | Placebo | TV-1106
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Early termination of study by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TV-1106 | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (12.86) | 56.4 (17.70) | 53.4 (15.66)
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 1 | 1 | 2
  >=40 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 7 | 12
  Missing | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 80.963 (24.1867) | 80.448 (13.3406) | 80.669 (17.9137)
Height [Mean (Standard Deviation); unit: cm] | 175.093 (9.1702) | 170.130 (8.5363) | 172.257 (8.8362)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.040 (6.1675) | 27.716 (3.3512) | 26.998 (4.6280)
Insulin-like Growth Factor 1 Standard Deviation Score [Mean (Standard Deviation); unit: standard deviations] — IGF-1 SDS represents the standard deviation from a 'normal' population.
  standard deviations | -2.00 (0.978) | -1.40 (0.545) | -1.66 (0.789)
Duration of Growth-Hormone Deficiency Diagnosis [Mean (Standard Deviation); unit: years] | 9.270 (9.3120) | 11.104 (13.1631) | 10.318 (11.2932)
Growth-Hormone Deficiency Onset [Count of Participants; unit: Participants]
  Adult (>+18 years) | 5 | 7 | 12
  Childhood (<18 years) | 1 | 1 | 2
Cause of Growth-Hormone Deficiency [Count of Participants; unit: Participants]
  Secreting pituitary adenoma | 0 | 1 | 1
  Non-secreting pituitary adenoma | 3 | 2 | 5
  Idiopathic | 0 | 1 | 1
  Other | 3 | 4 | 7
Prior Treatment for Growth-Hormone Deficiency [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 3
  No | 0 | 0 | 0
  Missing | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Body Fat Mass at Baseline, Week 24 and Endpoint in Core Period
Description: The primary efficacy measure for the study was body fat mass (kg) measured by DXA imaging. The primary outcome as defined in the protocol was the change from baseline to week 24 in body fat mass. Due to the early termination of the study, observed values including endpoint values are reported. Endpoint is the last observed value.
Time Frame: Baseline (Day 1, pre-dose), Week 24, Endpoint in Core period
Population: ITT
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
kg
  Baseline | 24.38 (7.495) | 29.50 (10.922)
  Week 24: number analyzed (Participants) | 1 | 1
  Week 24 | 28.90 (NA) — Value from a single individual | 31.80 (NA) — Value from a single individual
  Endpoint: number analyzed (Participants) | 3 | 6
  Endpoint | 23.27 (7.389) | 31.05 (13.256)

2. Secondary Outcome: Total Trunk Fat at Baseline, Week 24 and Endpoint in Core Period
Description: Trunk fat (kg) was assessed based on DXA results. Trunk fat was defined as fat mass - (total arm fat + total leg fat + total head fat). The outcome as defined in the protocol was the within-patient change from baseline to week 24 in trunk fat. Due to the early termination of the study, observed values including endpoint values are reported. Endpoint is the last observed value.
Time Frame: Baseline (Day 1, pre-dose), Week 24, Endpoint in Core Period
Population: ITT
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
kg
  Baseline | 12.02 (4.716) | 15.05 (5.041)
  Week 24: number analyzed (Participants) | 1 | 1
  Week 24 | 15.60 (NA) — Value from a single individual | 12.60 (NA) — Value from a single individual
  Endpoint: number analyzed (Participants) | 3 | 6
  Endpoint | 11.20 (4.173) | 15.05 (6.369)

3. Secondary Outcome: Insulin-Like Growth Factor 1 Standard Deviation Score (IGF-I SDS) at Baseline, Week 24 and Endpoint in Core Period
Description: IGF-I SDS, as reported by the central laboratory, was a key secondary variable. The week 24 value is a trough value as it was taken 7 days after the last TV-1106 or placebo injection. The outcome as defined in the protocol was the within-patient change from baseline to week 24. Due to the early termination of the study, observed values including endpoint values are reported. Endpoint is the last observed value and is of variable length of time since last TV-1106 or placebo injection.
Time Frame: Baseline (Day 1, pre-dose), Week 24, Endpoint in Core Period
Population: ITT
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
standard deviation score
  Baseline | -2.00 (0.978) | -1.40 (0.545)
  Week 24: number analyzed (Participants) | 1 | 1
  Week 24 | -2.00 (NA) — Value from a single individual | -1.30 (NA) — Value from a single individual
  Endpoint: number analyzed (Participants) | 5 | 6
  Endpoint | -1.66 (0.493) | -0.67 (0.896)

4. Secondary Outcome: Scored Analysis of Quality of Life Assessment of GH Deficiency in Adults (QoL-AGHDA) at Baseline, Week 24 and Endpoint in Core Period
Description: The AGHDA instrument is comprised of 25 questions, with yes or no answers. To each of the 25 questions comprising QOL AGHDA, a score of 1 was assigned if the answer was affirmative and 0 if the answer was negative. Data reported is the total score across the 25 questions for a total range of 0-25 with higher scores representing a poorer quality of life. The outcome as defined in the protocol was the within-patient change from baseline to week 24. Due to the early termination of the study, observed values including endpoint values are reported. Endpoint is the last observed value.
Time Frame: Baseline (Day 1, pre-dose), Week 24, Endpoint in Core Period
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
units on a scale
  Baseline | 3.8 (5.46) | 9.6 (8.14)
  Week 24: number analyzed (Participants) | 1 | 1
  Week 24 | 1.0 (NA) — Value from a single individual | 0.0 (NA) — Value from a single individual
  Endpoint | 2.8 (4.62) | 6.5 (6.12)

5. Secondary Outcome: Participants With Adverse Events During the Core Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents usual activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
Participants
  >=1 adverse event | 3 | 4
  Severe adverse event | 1 | 0
  Treatment-related adverse event | 0 | 2
  Deaths | 0 | 0
  Other serious adverse events | 1 | 0
  Discontinued from study drug due to adverse events | 1 | 0

6. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Blood and Urine Test Results
Description: Parameters with potentially clinically significant abnormal test results include - Serum chemistry: blood urea nitrogen, creatinine and bilirubin - Hematology: leukocytes, hemoglobin, hematocrit, platelets and neutrophils - Urinalysis: none Significance criteria are listed below with the test.
Time Frame: Day 1 up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
Participants
  Blood urea nitrogen: >=10.71 mmol/L | 0 | 1
  Creatinine: >=177 mmol/L | 0 | 1
  Bilirubin: >=34.2 mmol/L | 2 | 0
  Leukocytes: <=3.0 10^9/L | 1 | 0
  Hemoglobin: (male) <=115 g/L | 1 | 0
  Hematocrit: (male) <0.37 L/L | 1 | 0
  Platelets: <=75 10^9/L | 1 | 0
  Neutrophils: <=1.0 10^9/L | 1 | 0

7. Secondary Outcome: Shift From Baseline To Endpoint in Core Period in Electrocardiogram Findings
Description: Shifts represented as baseline - endpoint value (last observed post-baseline value). Abnormal NCS indicates an abnormal but not clinically significant finding. Abnormal CS indicates an abnormal and clinically significant finding.
Time Frame: Day 1 up to Week 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
Participants
  Normal - Normal | 4 | 6
  Normal - Abnormal NCS | 1 | 0
  Normal - Abnormal CS | 0 | 0
  Abnormal NCS - Normal | 1 | 1
  Abnormal NCS - Abnormal NCS | 0 | 1
  Abnormal NCS - Abnormal CS | 0 | 0

8. Secondary Outcome: Thyroid Stimulating Hormone (TSH) at Baseline and Endpoint
Description: One measure of changes in replacement hormones.
Time Frame: Baseline (Day 1, pre-dose), Endpoint (up to Week 24)
Population: Safety population of participants reporting data
Measure: Mean (Standard Deviation); unit: MIU/L
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
MIU/L
  Baseline: number analyzed (Participants) | 6 | 6
  Baseline | 0.365 (0.3791) | 1.028 (2.0259)
  Endpoint: number analyzed (Participants) | 6 | 7
  Endpoint | 0.545 (0.5439) | 0.796 (1.6971)

9. Secondary Outcome: Free Thyroxin (Free T4) at Baseline and Endpoint
Description: One measure of changes in replacement hormones.
Time Frame: Baseline (Day 1, pre-dose), Endpoint (up to Week 24)
Population: Safety population of participants reporting data
Measure: Mean (Standard Deviation); unit: PMOL/L
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
PMOL/L
  Baseline: number analyzed (Participants) | 6 | 7
  Baseline | 17.22 (5.375) | 15.26 (1.696)
  Endpoint | 15.65 (2.180) | 14.54 (3.259)

10. Secondary Outcome: Triiodothyronine (Total T3) at Baseline and Endpoint
Description: One measure of changes in replacement hormones.
Time Frame: Baseline (Day 1, pre-dose), Endpoint (up to Week 24)
Population: Safety population of participants reporting data
Measure: Mean (Standard Deviation); unit: NMOL/L
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
NMOL/L
  Baseline: number analyzed (Participants) | 6 | 7
  Baseline | 1.80 (1.228) | 1.71 (0.302)
  Endpoint: number analyzed (Participants) | 6 | 7
  Endpoint | 1.32 (0.133) | 1.64 (0.351)

11. Secondary Outcome: Glycated Hemoglobin (HbA1c) at Baseline and Endpoint
Description: One measure of glucose homeostasis.
Time Frame: Baseline (Day 1, pre-dose), Endpoint (up to Week 24)
Population: Safety population of participants reporting data
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
percentage of total hemoglobin
  Baseline: number analyzed (Participants) | 6 | 7
  Baseline | 5.53 (0.647) | 5.49 (0.422)
  Endpoint: number analyzed (Participants) | 6 | 7
  Endpoint | 5.45 (0.797) | 5.51 (0.358)

12. Secondary Outcome: Fasting Blood Glucose at Baseline and Endpoint
Description: One measure of glucose homeostasis.
Time Frame: Baseline (Day 1, pre-dose), Endpoint (up to Week 24)
Population: Safety population of participants reporting data
Measure: Mean (Standard Deviation); unit: MMOL/L
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
MMOL/L
  Baseline | 5.37 (2.389) | 4.83 (0.320)
  Endpoint | 4.82 (0.818) | 5.01 (0.344)

13. Secondary Outcome: Insulin at Baseline and Endpoint
Description: One measure of glucose homeostasis.
Time Frame: Baseline (Day 1, pre-dose), Endpoint (up to Week 24)
Population: Safety population of participants reporting data
Measure: Mean (Standard Deviation); unit: PMOL/L
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
PMOL/L
  Baseline | 68.0 (68.90) | 57.0 (22.68)
  Endpoint: number analyzed (Participants) | 6 | 7
  Endpoint | 65.0 (49.68) | 94.3 (89.04)

14. Secondary Outcome: Local Tolerability Assessed by Injection Site Reactions
Description: Participants reporting at least one injection site reaction.
Time Frame: Daay 1 up to Week 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 6 | 8
Participants
  Pain: number analyzed (Participants) | 6 | 7
  Pain | 0 | 2
  Tenderness | 0 | 1
  Erythema: number analyzed (Participants) | 6 | 7
  Erythema | 0 | 0
  Warmth: number analyzed (Participants) | 6 | 7
  Warmth | 0 | 0
  Swelling: number analyzed (Participants) | 6 | 7
  Swelling | 0 | 0

15. Secondary Outcome: Pharmacokinetic Serum Concentration of TV1106 by Nominal Sampling Timepoints
Description: Weeks 4 and 8 serum samples obtained 2 days after TV1106 administration. Weeks 12 and 24 serum samples obtained 7 days after TV1106 administration. Week 16 serum samples obtained 1 day after TV1106 administration.
Time Frame: Baseline (Day 1, pre-dose), Weeks 4, 8, 12, 16, 24
Population: Safety population of participants treated with TV1106
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Placebo | TV-1106
Number analyzed (Participants) | 0 | 8
ng/mL
  Baseline |  | NA [0.0 to 0.0] — Only min/max values reported where > 50% of results are below the limit of quantitation.
  Week 4, Day 2: number analyzed (Participants) | 0 | 4
  Week 4, Day 2 |  | NA [0.0 to 5.8] — Only min/max values reported where > 50% of results are below the limit of quantitation.
  Week 8, Day 2: number analyzed (Participants) | 0 | 3
  Week 8, Day 2 |  | 4.50 [0.0 to 4.7]
  Week 12, Day 7: number analyzed (Participants) | 0 | 2
  Week 12, Day 7 |  | NA [0.0 to 0.0] — Only min/max values reported where > 50% of results are below the limit of quantitation.
  Week 16, Day 1: number analyzed (Participants) | 0 | 2
  Week 16, Day 1 |  | 9.05 [6.6 to 11.5]
  Week 24, Day 7: number analyzed (Participants) | 0 | 1
  Week 24, Day 7 |  | NA [0.0 to 0.0] — Only min/max values reported where > 50% of results are below the limit of quantitation.

ADVERSE EVENTS:
Time Frame: Core Period: Day 1 to Week 24 Extension Period: Week 25-26
Groups:
- Placebo - Core Period: Placebo was injected subcutaneously once weekly on the same day and time for 24 weeks during the Core Period. To maintain the blind, placebo could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 to match the effect of dose titration. Participants who completed the Core Period were eligible to enter an open-label extension phase for 12 additional months where all participants received treatment with TV-1106.
- TV-1106 - Core Period: TV-1106 was injected subcutaneously once weekly on the same day and time for 24 weeks during the Core Period. A common starting dose was 5.0 mg. Doses could be titrated by an unblinded central reader on weeks 4, 8, 12 and 16 until the participant's insulin-like growth factor 1 (IGF-1) standard deviation score (SDS) was within the range of -0.5 to +1.5. Participants who completed the Core Period were eligible to enter an open-label extension phase for 12 additional months where all participants received treatment with TV-1106.
- TV-1106 - Extension Period: Participants from both the Placebo and TV-1106 groups who completed the Core Period were eligible to enter an open-label extension phase for 12 additional months where all participants received treatment with TV-1106. Due to early termination of the study, two participants spent a maximum of two weeks in the extension period.
Arm/Group | Placebo - Core Period | TV-1106 - Core Period | TV-1106 - Extension Period
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 3/6 | 4/8 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Core Period (N=6) | TV-1106 - Core Period (N=8) | TV-1106 - Extension Period (N=2)
Pituitary haemorrhage (Endocrine disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Core Period (N=6) | TV-1106 - Core Period (N=8) | TV-1106 - Extension Period (N=2)
Injection site pain (General disorders) | 0 | 2 (2) | 0
Injection site swelling (General disorders) | 0 | 0 | 1 (2)
Injection site rash (General disorders) | 0 | 0 | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 (1) | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 (1) | 0
Haematuria (Renal and urinary disorders) | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.